CLINICAL TRIAL: NCT05583461
Title: Ventilator-induced Right Ventricular Injury During Electrical Impedance Tomography-based Positive End-expiratory Pressure Titration in Patients With Acute Respiratory Distress Syndrome: a Pilot Physiological Study.
Brief Title: Ventilator-induced Right Ventricular Injury During EIT-based PEEP Titration in Patients With ARDS
Acronym: RIGHTENARDS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Tommaso Pettenuzzo, MD, University of Padova
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 5546/AO/22
Record Dates: First submitted 2022-10-13; First posted 2022-10-17 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Acute Respiratory Distress Syndrome; Right Ventricular Dysfunction
Keywords: Acute respiratory distress syndrome; Mechanical ventilation; Right ventricular dysfunction; Positive end-expiratory pressure; Electrical impedance tomography; Echocardiography
MeSH Terms: conditions — Respiratory Distress Syndrome; Ventricular Dysfunction, Right

STUDY DESIGN:
Intervention Model Description: Randomized sequence of application of four levels of positive end-expiratory pressure in adult patients requiring invasive controlled mechanical ventilation for acute respiratory distress syndrome
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Being sedated and paralyzed, included patients will not be aware of the study phase.
  The investigators performing the echocardiographic exams will be blinded to the experimental setting because the PEEP level set at the ventilator will be covered.
  The echocardiographic measurement will be performed offline with no information on the experimental settings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PEEP level according to the low PEEP-FiO2 table (Experimental): Positive end-expiratory pressure (PEEP) level selected based on patient's fraction of inspired oxygen (FiO2) according to the low PEEP-FiO2 table proposed by the Acute Respiratory Distress Syndrome Network Guidelines
  Interventions: Procedure: Positive end-expiratory pressure titration
- PEEP minimizing the risk of overdistension and atelectasis (Experimental): Positive end-expiratory pressure (PEEP) level selected based on the intersection between the curves of the cumulative percentages of compliance loss due to alveolar overdistension and atelectasis, respectively, as assessed with an electrical impedance tomography-based decremental PEEP trial
  Interventions: Procedure: Positive end-expiratory pressure titration
- PEEP minimizing the risk of overdistension (Experimental): Highest positive end-expiratory pressure (PEEP) level associated with no alveolar overdistention selected based on the curve of the cumulative percentage of compliance loss due to alveolar overdistension, as assessed with an electrical impedance tomography-based decremental PEEP trial
  Interventions: Procedure: Positive end-expiratory pressure titration
- PEEP minimizing the risk of atelectasis (Experimental): Lowest positive end-expiratory pressure (PEEP) level associated with no alveolar collapse selected based on the curve of the cumulative percentage of compliance loss due to alveolar collapse, as assessed with an electrical impedance tomography-based decremental PEEP trial
  Interventions: Procedure: Positive end-expiratory pressure titration

INTERVENTIONS:
Procedure: Positive end-expiratory pressure titration — Positive end-expiratory pressure level

SUMMARY:
Right ventricular failure may be associated with mortality in patients with acute respiratory distress syndrome (ARDS). Mechanical ventilation may promote right ventricular failure by inducing alveolar overdistention and atelectasis. Electrical impedance tomography (EIT) is a bedside non-invasive technique assessing the regional distribution of lung ventilation, thus helping titrating positive end-expiratory pressure (PEEP) to target the minimum levels of alveolar overdistension and atelectasis. The aim of this physiologic randomized crossover trial is to assess right ventricular size and function with transthoracic echocardiography with different levels of PEEP in adult patients with moderate-to-severe ARDS undergoing controlled invasive mechanical ventilation: the level of PEEP determined according to the ARDS Network low PEEP-FiO2 table, the PEEP value that minimizes the risk of alveolar overdistension and atelectasis (as determined by EIT), the highest PEEP value minimizing the risk of alveolar overdistension (as determined by EIT), and the lowest PEEP level that minimizes the risk of alveolar atelectasis (as determined by EIT). Our findings may offer valuable insights into the level of PEEP favoring right ventricular protection during mechanical ventilation in patients with ARDS.

DETAILED DESCRIPTION:
Acute respiratory distress syndrome (ARDS) is a diffuse pulmonary inflammatory disease with multifactorial etiology that is very common in patients admitted to the intensive care unit (ICU) and is associated with unsatisfactory short- and long-term prognosis. Patients with ARDS can develop right ventricular (RV) failure, which occurs in 22-50% of patients despite lung protective ventilation and is associated with increased mortality. Despite being required to ensure survival of patients with ARDS, mechanical ventilation itself may have injurious effects on RV function. First, high transpulmonary pressure, secondary to the use of high tidal volume, plateau pressure or positive end-expiratory pressure (PEEP), can cause alveolar overdistension, especially in the aerated parenchymal regions, and collapse of alveolar vessels. The consequent increase in pulmonary arterial pressure may lead to excessively high RV afterload and reduced systolic function. Second, the development of parenchymal atelectasis potentially secondary to the application of low tidal volumes and/or PEEP may increase pulmonary vascular resistance because of extra-alveolar vascular collapse. Finally, mechanical ventilation can have indirect effects on pulmonary circulation and RV function, mediated by alveolar oxygenation, acidosis, and hypercapnia.

The application of PEEP can prevent cyclic opening and closing of the alveoli (i.e., atelectrauma) and improve oxygenation. Ideally, PEEP should maintain lung recruitment and optimize oxygenation and dead space, while at the same time avoiding alveolar overdistension and hemodynamic complications. However, the PEEP titration strategy in patients with ARDS is still widely debated, due to the variability of the effects of PEEP in different patients and different lung parenchymal regions in the same patient. Depending on the extent of potentially recruitable lung parenchyma and the distribution of lung damage, the application of PEEP can cause alveolar overdistension and promote RV failure and/or favor alveolar recruitment and improve RV function. Therefore, it is stil unclear what level of PEEP is associated with the optimization of RV function in patients with ARDS. We may hypothesize that the level of PEEP able to reduce alveolar collapse without increasing overdistension may improve RV function.

Several strategies have been suggested to assess lung recruitability and PEEP responsiveness in patients with ARDS. Electrical impedance tomography (EIT) is a bedside non-invasive technique that monitors the regional distribution of lung ventilation. The choice of the PEEP value that minimizes the extent of overdistension and atelectasis, as assessed with EIT, was associated with better respiratory mechanics and survival in patients with severe ARDS in some pilot studies.

The aim of this prospective pathophysiological interventional study is to evaluate the variation of RV size and function with transthoracic echocardiography in adult patients requiring invasive controlled mechanical ventilation for moderate-to-severe ARDS with four different PEEP values applied according to a randomized sequence in each patient:

* The level of PEEP determined according to the ARDS Network low PEEP-fraction of inspired oxygen (FiO2) table;
* The PEEP value that minimizes the risk of overdistension and atelectasis, as determined by EIT;
* The highest PEEP value that minimizes the risk of overdistension, as determined by EIT;
* The lowest PEEP level that minimizes the risk of atelectasis, as determined by EIT.

The primary hypothesis of the study is that the level of PEEP that simultaneously minimizes alveolar overdistension and collapse is associated with better RV function than the PEEP level selected based on the low PEEP-FiO2 table and PEEP levels that minimize overdistension and collapse, separately. The secondary hypotheses of the study are that: 1) the level of PEEP that minimizes overdistension is associated with better RV function than the level of PEEP that minimizes collapse; 2) the PEEP level that minimizes alveolar collapse is associated with greater pulmonary air content, as assessed by lung ultrasound, compared to the PEEP levels chosen based on the low PEEP-FiO2 table, the PEEP level that minimizes overdistension and collapse simultaneously, and the PEEP level that minimizes overdistension.

The physiological data obtained from this study may offer valuable insights into the right ventricular-protective level of PEEP in patients with ARDS and support future large randomized studies investigating PEEP levels associated with improved patient survival.

ELIGIBILITY:
Inclusion criteria:

1. Moderate to severe acute respiratory distress syndrome
2. Inclusion within 72 hours of acute respiratory distress syndrome diagnosis
3. Endotracheal intubation or tracheostomy

Exclusion criteria:

1. Age lower than 18 years old
2. Pregnancy
3. Absence of informed consent
4. Thoracic surgery or lung transplant during the admission
5. Contraindications to recruitment maneuvers (mean arterial pressure lower than 65 mmHg despite administration of fluids or vasopressors, active air leaks through a chest tube, pneumothorax or subcutaneous or mediastinal emphysema in absence of chest drainage)
6. Contraindications to electrical impedance tomography (contraindication to recruitment maneuvers, presence of pacemakers or other electronic devices in the chest, injuries or burns in the electrode placement area)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Right ventricle diameter 1 | Measured after 20 minutes from the application of each of the four levels of PEEP
  Maximal transversal dimension in the basal one third of right ventricular inflow at end-diastole in the right ventricle-focused apical four-chamber view
Right ventricle diameter 2 | Measured after 20 minutes from the application of each of the four levels of PEEP
  Transversal right ventricular diameter in the middle third of right ventricular inflow, approximately halfway between the maximal basal diameter and the apex, at the level of papillary muscles at end-diastole.
Right ventricle fractional area change | Measured after 20 minutes from the application of each of the four levels of PEEP
  Ratio of the difference between end-diastolic area and end-systolic area to end-diastolic area, which are determined after manual tracing of right ventricular endocardial border from the lateral tricuspid annulus along the free wall to the apex and back to medial tricuspid annulus, along the interventricular septum at end-diastole and at end-systole, in the right ventricle-focused apical four-chamber view
Eccentricity index | Measured after 20 minutes from the application of each of the four levels of PEEP
  Ratio between two left ventricular axes, one parallel to the interventricular septum and one perpendicular to this, in the mid-papillary parasternal short axis view
Tricuspid annular plane systolic excursion | Measured after 20 minutes from the application of each of the four levels of PEEP
  Tricuspid annular longitudinal excursion by M-mode, measured between end-diastole and peak systole in the apical four-chamber view that achieves parallel alignment of Doppler beam with right ventricular free wall longitudinal excursion
Systolic velocity of the lateral tricuspid annulus derived from tissue Doppler imaging | Measured after 20 minutes from the application of each of the four levels of PEEP
  Peak systolic velocity of lateral tricuspid annulus by pulsed-wave tissue Doppler imaging in the apical four-chamber view that achieves parallel alignment of Doppler beam with right ventricular free wall longitudinal excursion
Right ventricular index of myocardial performance | Measured after 20 minutes from the application of each of the four levels of PEEP
  The ratio of the sum between isovolumic contraction and relaxation times to ejection time measured by pulsed-wave tissue Doppler imaging in the apical four-chamber view that achieves parallel alignment of Doppler beam with right ventricular free wall longitudinal excursion
Right ventricle systolic pressure | Measured after 20 minutes from the application of each of the four levels of PEEP
  Calculated from the velocity of tricuspid regurgitation jet, measured in the view allowing the highest value, by applying simplified Bernoulli equation and adding right atrial pressure estimated from central venous pressure
Myocardial isovolumic acceleration | Measured after 20 minutes from the application of each of the four levels of PEEP
  Ratio of lateral tricuspid annulus peak velocity during isovolumic contraction to acceleration time by pulsed-wave tissue Doppler imaging in the apical four-chamber view that achieves parallel alignment of Doppler beam with right ventricular free wall longitudinal excursion
Right ventricle stroke index | Measured after 20 minutes from the application of each of the four levels of PEEP
  Ratio of right ventricular stroke volume, calculated as product between velocity-time integral at the level of pulmonary valve and transverse area of right ventricular outflow tract in the aortic valve-level parasternal short axis view during systole, and body surface area
Right ventricle stroke work index | Measured after 20 minutes from the application of each of the four levels of PEEP
  Product between right ventricle stroke index and right ventricle systolic pressure
Right ventricular free wall longitudinal strain | Measured after 20 minutes from the application of each of the four levels of PEEP
  Peak value of longitudinal speckle-tracking-derived strain, averaged over the three segments of the right ventricular free wall, after manual tracing of right ventricular endocardial border from the lateral tricuspid annulus along the free wall to the apex and back to medial tricuspid annulus in right ventricle-focused apical four-chamber view

SECONDARY OUTCOMES:
Ventilator settings | Measured after 20 minutes from the application of each of the four levels of PEEP
  Tidal volume, respiratory rate, fraction of inspired oxygen, inspiratory to expiratory time
Respiratory mechanics | Measured after 20 minutes from the application of each of the four levels of PEEP
  Plateau pressure, total positive end-expiratory pressure, driving pressure, mechanical power
Arterial blood gas analysis | Measured after 20 minutes from the application of each of the four levels of PEEP
  pH, arterial partial pressure of carbon dioxide, arterial partial pressure of oxygen, arterial oxygen saturation, bicarbonate, lactate
Dead space | Measured after 20 minutes from the application of each of the four levels of PEEP
  Estimated from the Bohr-Enghoff equation (ratio of the difference between arterial partial pressure of carbon dioxide and end-tidal carbon dioxide to arterial partial pressure of carbon dioxide)
Ventilatory ratio | Measured after 20 minutes from the application of each of the four levels of PEEP
  Product between minute ventilation and arterial partial pressure of carbon dioxide, divided by predicted body weight x 100 x 37.5
Shunt | Measured after 20 minutes from the application of the intervention
  Calculated as (1 - arterial oxygen saturation) divided by (1 - central venous oxygen saturation)
Hemodynamics | Measured after 20 minutes from the application of the intervention
  Systolic blood pressure, diastolic blood pressure, mean arterial pressure, heart rate, central venous pressure, dosage of vasoactive agents
Pleural and lung ultrasound | Measured after 20 minutes from the application of the intervention
  Lung ultrasound score, lung reaeration score
Renal ultrasound | Measured after 20 minutes from the application of the intervention
  Renal resistive index, renal venous stasis index
Ultrasound image quality | Measured after 20 minutes from the application of the intervention
  Quality assessed according to the 2018 American College of Emergency Physicians Guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Tommaso Pettenuzzo, MD, Principal Investigator — Institute of Anesthesiology and Intensive Care, Padova University Hospital
Locations (1):
- University Hospital of Padua, Padua, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fan E, Brodie D, Slutsky AS. Acute Respiratory Distress Syndrome: Advances in Diagnosis and Treatment. JAMA. 2018 Feb 20;319(7):698-710. doi: 10.1001/jama.2017.21907. PMID 29466596
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Background] Gattinoni L, Marini JJ, Pesenti A, Quintel M, Mancebo J, Brochard L. The "baby lung" became an adult. Intensive Care Med. 2016 May;42(5):663-673. doi: 10.1007/s00134-015-4200-8. Epub 2016 Jan 18. PMID 26781952
- [Background] Bellani G, Laffey JG, Pham T, Fan E, Brochard L, Esteban A, Gattinoni L, van Haren F, Larsson A, McAuley DF, Ranieri M, Rubenfeld G, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Epidemiology, Patterns of Care, and Mortality for Patients With Acute Respiratory Distress Syndrome in Intensive Care Units in 50 Countries. JAMA. 2016 Feb 23;315(8):788-800. doi: 10.1001/jama.2016.0291. PMID 26903337
- [Background] Bein T, Grasso S, Moerer O, Quintel M, Guerin C, Deja M, Brondani A, Mehta S. The standard of care of patients with ARDS: ventilatory settings and rescue therapies for refractory hypoxemia. Intensive Care Med. 2016 May;42(5):699-711. doi: 10.1007/s00134-016-4325-4. Epub 2016 Apr 4. PMID 27040102
- [Background] Herridge MS, Tansey CM, Matte A, Tomlinson G, Diaz-Granados N, Cooper A, Guest CB, Mazer CD, Mehta S, Stewart TE, Kudlow P, Cook D, Slutsky AS, Cheung AM; Canadian Critical Care Trials Group. Functional disability 5 years after acute respiratory distress syndrome. N Engl J Med. 2011 Apr 7;364(14):1293-304. doi: 10.1056/NEJMoa1011802. PMID 21470008
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] Guerin C, Reignier J, Richard JC, Beuret P, Gacouin A, Boulain T, Mercier E, Badet M, Mercat A, Baudin O, Clavel M, Chatellier D, Jaber S, Rosselli S, Mancebo J, Sirodot M, Hilbert G, Bengler C, Richecoeur J, Gainnier M, Bayle F, Bourdin G, Leray V, Girard R, Baboi L, Ayzac L; PROSEVA Study Group. Prone positioning in severe acute respiratory distress syndrome. N Engl J Med. 2013 Jun 6;368(23):2159-68. doi: 10.1056/NEJMoa1214103. Epub 2013 May 20. PMID 23688302
- [Background] Papazian L, Forel JM, Gacouin A, Penot-Ragon C, Perrin G, Loundou A, Jaber S, Arnal JM, Perez D, Seghboyan JM, Constantin JM, Courant P, Lefrant JY, Guerin C, Prat G, Morange S, Roch A; ACURASYS Study Investigators. Neuromuscular blockers in early acute respiratory distress syndrome. N Engl J Med. 2010 Sep 16;363(12):1107-16. doi: 10.1056/NEJMoa1005372. PMID 20843245
- [Background] Tremblay LN, Slutsky AS. Ventilator-induced lung injury: from the bench to the bedside. Intensive Care Med. 2006 Jan;32(1):24-33. doi: 10.1007/s00134-005-2817-8. Epub 2005 Oct 18. No abstract available. PMID 16231069
- [Background] Kuipers MT, van der Poll T, Schultz MJ, Wieland CW. Bench-to-bedside review: Damage-associated molecular patterns in the onset of ventilator-induced lung injury. Crit Care. 2011;15(6):235. doi: 10.1186/cc10437. Epub 2011 Nov 30. PMID 22216838
- [Background] Slutsky AS, Ranieri VM. Ventilator-induced lung injury. N Engl J Med. 2013 Nov 28;369(22):2126-36. doi: 10.1056/NEJMra1208707. No abstract available. PMID 24283226
- [Background] Del Sorbo L, Slutsky AS. Acute respiratory distress syndrome and multiple organ failure. Curr Opin Crit Care. 2011 Feb;17(1):1-6. doi: 10.1097/MCC.0b013e3283427295. PMID 21157315
- [Background] Cressoni M, Cadringher P, Chiurazzi C, Amini M, Gallazzi E, Marino A, Brioni M, Carlesso E, Chiumello D, Quintel M, Bugedo G, Gattinoni L. Lung inhomogeneity in patients with acute respiratory distress syndrome. Am J Respir Crit Care Med. 2014 Jan 15;189(2):149-58. doi: 10.1164/rccm.201308-1567OC. PMID 24261322
- [Background] Yoshida T, Fujino Y, Amato MB, Kavanagh BP. Fifty Years of Research in ARDS. Spontaneous Breathing during Mechanical Ventilation. Risks, Mechanisms, and Management. Am J Respir Crit Care Med. 2017 Apr 15;195(8):985-992. doi: 10.1164/rccm.201604-0748CP. PMID 27786562
- [Background] Amato MB, Meade MO, Slutsky AS, Brochard L, Costa EL, Schoenfeld DA, Stewart TE, Briel M, Talmor D, Mercat A, Richard JC, Carvalho CR, Brower RG. Driving pressure and survival in the acute respiratory distress syndrome. N Engl J Med. 2015 Feb 19;372(8):747-55. doi: 10.1056/NEJMsa1410639. PMID 25693014
- [Background] Gattinoni L, Pelosi P, Crotti S, Valenza F. Effects of positive end-expiratory pressure on regional distribution of tidal volume and recruitment in adult respiratory distress syndrome. Am J Respir Crit Care Med. 1995 Jun;151(6):1807-14. doi: 10.1164/ajrccm.151.6.7767524.
- [Background] Santa Cruz R, Rojas JI, Nervi R, Heredia R, Ciapponi A. High versus low positive end-expiratory pressure (PEEP) levels for mechanically ventilated adult patients with acute lung injury and acute respiratory distress syndrome. Cochrane Database Syst Rev. 2013 Jun 6;2013(6):CD009098. doi: 10.1002/14651858.CD009098.pub2. PMID 23740697
- [Background] Carpenter TC, Stenmark KR. Hypoxia decreases lung neprilysin expression and increases pulmonary vascular leak. Am J Physiol Lung Cell Mol Physiol. 2001 Oct;281(4):L941-8. doi: 10.1152/ajplung.2001.281.4.L941. PMID 11557598
- [Background] Madjdpour C, Jewell UR, Kneller S, Ziegler U, Schwendener R, Booy C, Klausli L, Pasch T, Schimmer RC, Beck-Schimmer B. Decreased alveolar oxygen induces lung inflammation. Am J Physiol Lung Cell Mol Physiol. 2003 Feb;284(2):L360-7. doi: 10.1152/ajplung.00158.2002. Epub 2002 Oct 11. PMID 12388372
- [Background] Mekontso Dessap A, Voiriot G, Zhou T, Marcos E, Dudek SM, Jacobson JR, Machado R, Adnot S, Brochard L, Maitre B, Garcia JG. Conflicting physiological and genomic cardiopulmonary effects of recruitment maneuvers in murine acute lung injury. Am J Respir Cell Mol Biol. 2012 Apr;46(4):541-50. doi: 10.1165/rcmb.2011-0306OC. Epub 2011 Dec 1. PMID 22135358
- [Background] Vieillard-Baron A, Matthay M, Teboul JL, Bein T, Schultz M, Magder S, Marini JJ. Experts' opinion on management of hemodynamics in ARDS patients: focus on the effects of mechanical ventilation. Intensive Care Med. 2016 May;42(5):739-749. doi: 10.1007/s00134-016-4326-3. Epub 2016 Apr 1. PMID 27038480
- [Background] Fan E, Del Sorbo L, Goligher EC, Hodgson CL, Munshi L, Walkey AJ, Adhikari NKJ, Amato MBP, Branson R, Brower RG, Ferguson ND, Gajic O, Gattinoni L, Hess D, Mancebo J, Meade MO, McAuley DF, Pesenti A, Ranieri VM, Rubenfeld GD, Rubin E, Seckel M, Slutsky AS, Talmor D, Thompson BT, Wunsch H, Uleryk E, Brozek J, Brochard LJ; American Thoracic Society, European Society of Intensive Care Medicine, and Society of Critical Care Medicine. An Official American Thoracic Society/European Society of Intensive Care Medicine/Society of Critical Care Medicine Clinical Practice Guideline: Mechanical Ventilation in Adult Patients with Acute Respiratory Distress Syndrome. Am J Respir Crit Care Med. 2017 May 1;195(9):1253-1263. doi: 10.1164/rccm.201703-0548ST. PMID 28459336
- [Background] Gattinoni L, Caironi P, Cressoni M, Chiumello D, Ranieri VM, Quintel M, Russo S, Patroniti N, Cornejo R, Bugedo G. Lung recruitment in patients with the acute respiratory distress syndrome. N Engl J Med. 2006 Apr 27;354(17):1775-86. doi: 10.1056/NEJMoa052052. PMID 16641394
- [Background] Gattinoni L, Marini JJ. In search of the Holy Grail: identifying the best PEEP in ventilated patients. Intensive Care Med. 2022 Jun;48(6):728-731. doi: 10.1007/s00134-022-06698-x. Epub 2022 May 5. No abstract available. PMID 35513707
- [Background] Repesse X, Charron C, Vieillard-Baron A. Acute respiratory distress syndrome: the heart side of the moon. Curr Opin Crit Care. 2016 Feb;22(1):38-44. doi: 10.1097/MCC.0000000000000267. PMID 26627538
- [Background] Zochios V, Parhar K, Tunnicliffe W, Roscoe A, Gao F. The Right Ventricle in ARDS. Chest. 2017 Jul;152(1):181-193. doi: 10.1016/j.chest.2017.02.019. Epub 2017 Mar 4. PMID 28267435
- [Background] Schmitt JM, Vieillard-Baron A, Augarde R, Prin S, Page B, Jardin F. Positive end-expiratory pressure titration in acute respiratory distress syndrome patients: impact on right ventricular outflow impedance evaluated by pulmonary artery Doppler flow velocity measurements. Crit Care Med. 2001 Jun;29(6):1154-8. doi: 10.1097/00003246-200106000-00012. PMID 11395592
- [Background] Suter PM, Fairley B, Isenberg MD. Optimum end-expiratory airway pressure in patients with acute pulmonary failure. N Engl J Med. 1975 Feb 6;292(6):284-9. doi: 10.1056/NEJM197502062920604. PMID 234174
- [Background] Zochios V, Yusuff H, Schmidt M; Protecting the Right Ventricle Network (PRORVnet). Acute right ventricular injury phenotyping in ARDS. Intensive Care Med. 2023 Jan;49(1):99-102. doi: 10.1007/s00134-022-06904-w. Epub 2022 Oct 11. No abstract available. PMID 36219228
- [Background] Zapol WM, Snider MT. Pulmonary hypertension in severe acute respiratory failure. N Engl J Med. 1977 Mar 3;296(9):476-80. doi: 10.1056/NEJM197703032960903. PMID 834225
- [Background] Sato R, Dugar S, Cheungpasitporn W, Schleicher M, Collier P, Vallabhajosyula S, Duggal A. The impact of right ventricular injury on the mortality in patients with acute respiratory distress syndrome: a systematic review and meta-analysis. Crit Care. 2021 May 21;25(1):172. doi: 10.1186/s13054-021-03591-9. PMID 34020703
- [Background] Mekontso Dessap A, Boissier F, Charron C, Begot E, Repesse X, Legras A, Brun-Buisson C, Vignon P, Vieillard-Baron A. Acute cor pulmonale during protective ventilation for acute respiratory distress syndrome: prevalence, predictors, and clinical impact. Intensive Care Med. 2016 May;42(5):862-870. doi: 10.1007/s00134-015-4141-2. Epub 2015 Dec 9. PMID 26650055
- [Background] Lemarie J, Maigrat CH, Kimmoun A, Dumont N, Bollaert PE, Selton-Suty C, Gibot S, Huttin O. Feasibility, reproducibility and diagnostic usefulness of right ventricular strain by 2-dimensional speckle-tracking echocardiography in ARDS patients: the ARD strain study. Ann Intensive Care. 2020 Feb 13;10(1):24. doi: 10.1186/s13613-020-0636-2. PMID 32056017
- [Background] Volpicelli G, Elbarbary M, Blaivas M, Lichtenstein DA, Mathis G, Kirkpatrick AW, Melniker L, Gargani L, Noble VE, Via G, Dean A, Tsung JW, Soldati G, Copetti R, Bouhemad B, Reissig A, Agricola E, Rouby JJ, Arbelot C, Liteplo A, Sargsyan A, Silva F, Hoppmann R, Breitkreutz R, Seibel A, Neri L, Storti E, Petrovic T; International Liaison Committee on Lung Ultrasound (ILC-LUS) for International Consensus Conference on Lung Ultrasound (ICC-LUS). International evidence-based recommendations for point-of-care lung ultrasound. Intensive Care Med. 2012 Apr;38(4):577-91. doi: 10.1007/s00134-012-2513-4. Epub 2012 Mar 6. PMID 22392031
- [Background] Quisi A, Harbalioglu H, Ozel MA, Alici G, Genc O, Kurt IH. The association between the renal resistive index and the myocardial performance index in the general population. Echocardiography. 2020 Sep;37(9):1399-1405. doi: 10.1111/echo.14702. Epub 2020 Aug 10. PMID 32777128
- [Background] Husain-Syed F, Birk HW, Ronco C, Schormann T, Tello K, Richter MJ, Wilhelm J, Sommer N, Steyerberg E, Bauer P, Walmrath HD, Seeger W, McCullough PA, Gall H, Ghofrani HA. Doppler-Derived Renal Venous Stasis Index in the Prognosis of Right Heart Failure. J Am Heart Assoc. 2019 Nov 5;8(21):e013584. doi: 10.1161/JAHA.119.013584. Epub 2019 Oct 19. PMID 31630601
- [Background] Sella N, Pettenuzzo T, Zarantonello F, Andreatta G, De Cassai A, Schiavolin C, Simoni C, Pasin L, Boscolo A, Navalesi P. Electrical impedance tomography: A compass for the safe route to optimal PEEP. Respir Med. 2021 Oct;187:106555. doi: 10.1016/j.rmed.2021.106555. Epub 2021 Jul 30. PMID 34352563
- [Background] Chiumello D, Gotti M, Guanziroli M, Formenti P, Umbrello M, Pasticci I, Mistraletti G, Busana M. Bedside calculation of mechanical power during volume- and pressure-controlled mechanical ventilation. Crit Care. 2020 Jul 11;24(1):417. doi: 10.1186/s13054-020-03116-w. PMID 32653011
- [Background] Sinha P, Calfee CS, Beitler JR, Soni N, Ho K, Matthay MA, Kallet RH. Physiologic Analysis and Clinical Performance of the Ventilatory Ratio in Acute Respiratory Distress Syndrome. Am J Respir Crit Care Med. 2019 Feb 1;199(3):333-341. doi: 10.1164/rccm.201804-0692OC. PMID 30211618
- [Background] Rudski LG, Lai WW, Afilalo J, Hua L, Handschumacher MD, Chandrasekaran K, Solomon SD, Louie EK, Schiller NB. Guidelines for the echocardiographic assessment of the right heart in adults: a report from the American Society of Echocardiography endorsed by the European Association of Echocardiography, a registered branch of the European Society of Cardiology, and the Canadian Society of Echocardiography. J Am Soc Echocardiogr. 2010 Jul;23(7):685-713; quiz 786-8. doi: 10.1016/j.echo.2010.05.010. No abstract available. PMID 20620859
- [Background] Lang RM, Badano LP, Mor-Avi V, Afilalo J, Armstrong A, Ernande L, Flachskampf FA, Foster E, Goldstein SA, Kuznetsova T, Lancellotti P, Muraru D, Picard MH, Rietzschel ER, Rudski L, Spencer KT, Tsang W, Voigt JU. Recommendations for cardiac chamber quantification by echocardiography in adults: an update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. J Am Soc Echocardiogr. 2015 Jan;28(1):1-39.e14. doi: 10.1016/j.echo.2014.10.003. PMID 25559473
- [Background] American College of Emergency Physicians 2018 Guidelines. Accessible from www.acep.org.